CLINICAL TRIAL: NCT02762942
Title: Prospective Randomized Clinical Trial Comparing the Effect of Vaginal Misoprostol Synchronously With Supracervical Balloon Versus Vaginal Misoprostol Alone for Induction of Labor
Brief Title: Comparison of Vaginal Misoprostol Plus Supracervical Balloon Versus Vaginal Misoprostol Alone for Induction of Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Dra Angels Vives Argilagós, Obstetrician, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-002061-29; 2015-002061-29 (EudraCT Number)
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Induction of Labor; Cervical Ripening; Pregnancy
Keywords: cervical ripening; misoprostol; supracervical balloon; Foley catheter
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal misoprostol alone (Active Comparator): Women in this group will receive 25mcg of vaginal misoprostol every 4 hours up to a maximum of 5 doses. Misoprostol will be stopped in case of a favorable cervix or if the patient is in active labor. In case of no progression after 5 doses of misoprostol, intravenous oxytocin will be perfused 4 hours after the last dose of misoprostol according to local protocols
  Interventions: Drug: Misoprostol
- Vaginal misoprostol + Foley catheter (Experimental): Women in this group will receive 25mcg of vaginal misoprostol every 4 hours up to a maximum of 5 doses. At the same time a 16French Foley catheter will be inserted through the internal os with visualization of the cervix by sterile speculum examination. The catheter balloon will be inflated with 30 ml of sterile normal saline solution and then the catheter will be taped with gentle traction to the inner thigh of the patient until spontaneous expulsion. If this does not occur, the catheter will be deflated and removed after 12 hours. Misoprostol will be stopped in case of a favorable cervix or if the patient is in active labor. In case of no progression after 5 doses of misoprostol, intravenous oxytocin will be perfused 4 hours after the last dose of misoprostol.
  Interventions: Drug: Misoprostol; Device: Foley catheter

INTERVENTIONS:
Drug: Misoprostol — Administration of 25 mcg of vaginal misoprostol every 4 hours up to 5 doses
  Other Names: Misofar
Device: Foley catheter — Insertion of a Foley catheter (16French) through the internal os for a maximum of 12 hours
  Other Names: Supracervical balloon
  Arms: Vaginal misoprostol + Foley catheter

SUMMARY:
Demonstrate that with concomitant and synchronous use of supracervical balloon and vaginal misoprostol for induction of labour, vaginal delivery is achieved in less time compared with vaginal misoprostol alone.

ELIGIBILITY:
Inclusion criteria:

* Singleton pregnancy
* Cephalic presentation
* Reassuring fetal heart rate pattern
* Intact membranes
* Bishop score less than 6

Exclusion criteria

* Severe preeclampsia
* Prematurity ( < 37 weeks gestation dated by first trimester ultrasound)
* Previous cesarean section or previous uterine surgery
* Intrauterine growth restriction
* Premature rupture of membranes
* Maternal colonization with Streptococcus Agalactiae at any time during pregnancy
* Multifetal pregnancy
* Breech presentation
* Stillbirth
* Any contraindication for vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Induction to delivery time | 1 year

SECONDARY OUTCOMES:
Bishop score at 12 hours from the onset of induction | 1 year
Bishop score at 24 hours from the onset of induction | 1 year
Number of doses of misoprostol required | 1 year
Percentage of pregnant women requiring oxytocin | 1 year
Maximum dosage of oxytocin given (mU / min) | 1 year
Percentage of pregnant women requiring epidural analgesia | 1 year
Percentage of pregnant women with tachysystole and / or hypertonus with absence of fetal heart rate decelerations | 1 year
Percentage of pregnant women with tachysystole and / or hypertonus with fetal heart rate decelerations | 1 year
Percentage of pregnant women with intrapartum fever | 1 year
Percentage of pregnant women with maternal side effects | 1 year
Percentage of pregnant women with vaginal delivery within 12 hours from the onset of induction | 1 year
Percentage of pregnant women with vaginal delivery within 24 hours from the onset of induction | through study completion
Total rate of cesarean section | 1 year
Percentage of cesarean sections for failed induction | 1 year
Percentage of cesarean sections for nonreassuring fetal status | 1 year
Neonatal intensive care unit admission | 1 year
Apgar score at 5 minutes | 1 year
Umbilical artery ph | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Àngels Vives Argilagós, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264